CLINICAL TRIAL: NCT05937061
Title: Influence of Persistent Food Allergy on Nutritional Status of Children With Food Allergy
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: 20200133
Record Dates: First submitted 2023-04-05; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Milk allergy: Children with milk allergy.
  Interventions: Biological: Blood sample analysis; Radiation: Bone mineral density measurement (DXA); Other: Influence of food allergy on growth (intervention groups)
- Egg Allergy: Children with egg allergy
  Interventions: Biological: Blood sample analysis; Other: Anthropometrics measurement - at inclusion to the study (all groups).; Other: Influence of food allergy on growth (intervention groups)
- Peanut allergy: Children with peanut allergy
  Interventions: Biological: Blood sample analysis; Other: Anthropometrics measurement - at inclusion to the study (all groups).; Other: Influence of food allergy on growth (intervention groups)
- Control group: Patients withhout food allergy (bee venom or drug allergy).
  Interventions: Biological: Blood sample analysis; Other: Anthropometrics measurement - at inclusion to the study (all groups).

INTERVENTIONS:
Biological: Blood sample analysis — Analysis of complete blood count, hemogram, serum proteins, serum iron status (iron, transferin, ferritin). Group comparison - intervention vs. control.
Other: Anthropometrics measurement - at inclusion to the study (all groups). — Measurement of body height (cm), weight (kg) and calculating BMI (kg/m2). Group comparison - intervention vs. control.
  Groups: Control group; Egg Allergy; Peanut allergy
Radiation: Bone mineral density measurement (DXA) — Analysis of bone mineral density with DXA in patients with milk allegy. Analysis ordered by medical doctor.
  Groups: Milk allergy
Other: Influence of food allergy on growth (intervention groups) — Gathering the data about of body height (cm), weight (kg) BMI (kg/m2) at the diagnosis of food allergy and comparison versus data at the enrollment in the study to asses growth.
  Groups: Egg Allergy; Milk allergy; Peanut allergy

SUMMARY:
The goal of this single center retrospective cohort study with observational longitudinal follow up is to compare food - allergic children (egg, milk and peanut allergy) with children in control group (children without any food allergy).

The main question[s] it aims to answer are:

* If children with food allergy groups will have lower food intake od micronutrients?
* If growth in children with food allergy is worse as in control group?
* If they are more malnourished and in the food allergies group is more stunting than in the control group?
* If children with milk allergy have lower intake of calcium in their diet and lower mineral bone density?

Participants will be asked to do 3 day food diary and to have blood analysed (hemograme, complete blood count, serum iron status, serum protein).

If there is a comparison group: Researchers will compare milk, egg and peanut allergy group to the control group (peers without food allergy) to see if the food allergy affects growth, macronutrient, micronutrient intake.

DETAILED DESCRIPTION:
Study design A single center retrospective cohort study with observational longitudinal follow up will be performed. The study will include three intervention groups (milk, egg and peanut allergy) and a control group (children with no food allergy). Patients will be 2 to 12 years old. The patients will be recruited at our University Medical Center Ljubljana, Pediatric hospital Ljubljana, outpatient care of our Department for Allergology, Rheumatology and Clinical Immunology. This study will be conducted according to the guidelines in Declaration of Helsinki and approved by Ethics Committee of Slovenia. Written informed consent will be obtained from all the subject's caregivers. The investigators will follow patients from confirmation of food allergy on and will collect data about their weight (kg) and height (cm) from our information system or patients' doctor (or caregiver). The investigators will collect data prospectively for 3 months from outpatient registry of our clinic. At the day of appointment patients will bring 3-day nutrition diary which was later analyzed by dietitian. The parents will attend an appointment by the dietitian where they will be informed about food diary analysis result and given the advice to enhance nutrition if necessary.

ELIGIBILITY:
Inclusion Criteria:

* IgE-mediated food allergy (skin prick test and/or speciﬁc IgE combined with an allergy focused history)

Exclusion Criteria:

* other chronic diseases (except atopic dermatitis, asthma, anaphylactic reaction, angioedema),
* vegetarian or vegan nutrition.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with food-allergy were between 2 and 12 years old. All children in intervention group had IgE-mediated food allergy (skin prick test and/or speciﬁc IgE combined with an allergy focused history) to milk, egg or peanut.
  In control group there were children between 2 and 12 years old, with no food allergy (patients with bee venom or drug allergy).
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Influence of food allergy on growth | 6 years
  Patients body weight (kg), height (cm) and use WHO growth curves to asses their growth and nutritional status and compare the to control group. Comparison of their measurements against the measurements at the time od diagnosis to asses the influence on growth.
Influence of food allergy on food intake and nutrient intake | 29 months
  Patients caregivers will deliver 3 - day food diary and dietitan will analyse it (energy intake - kcals/KJ, intake of proteins kg/kg of body weight/day, intake of calcium and iron in mg/day and %of fat, %of carbohydrates and % of proteins in their nutrition. It will all be compared to the control group..
Influence of food allergy on blood sampling analysis | 29 months
  Blood sample analysis will be performed and results of intervention groups compared versus control group
Influence of milk allergy on bone mineral density | 29 months
  Data of bone mineral density will be gathered from our patients database and analysed

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Avcin, prof., Study Director — Head of Department of Clinical Immunology, Rheumatology and Allergology
Locations (1):
- Universitiy Medical center Ljubljana, division for Pediatrics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berni Canani R, Leone L, D'Auria E, Riva E, Nocerino R, Ruotolo S, Terrin G, Cosenza L, Di Costanzo M, Passariello A, Coruzzo A, Agostoni C, Giovannini M, Troncone R. The effects of dietary counseling on children with food allergy: a prospective, multicenter intervention study. J Acad Nutr Diet. 2014 Sep;114(9):1432-9. doi: 10.1016/j.jand.2014.03.018. Epub 2014 Jun 3. PMID 24933388
- [Background] Beck C, Koplin J, Dharmage S, Wake M, Gurrin L, McWilliam V, Tang M, Sun C, Foskey R, Allen KJ; HealthNuts Investigators. Persistent Food Allergy and Food Allergy Coexistent with Eczema Is Associated with Reduced Growth in the First 4 Years of Life. J Allergy Clin Immunol Pract. 2016 Mar-Apr;4(2):248-56.e3. doi: 10.1016/j.jaip.2015.08.009. Epub 2015 Oct 2. PMID 26441150
- [Background] Meyer R, De Koker C, Dziubak R, Godwin H, Dominguez-Ortega G, Chebar Lozinsky A, Skrapac AK, Gholmie Y, Reeve K, Shah N. The impact of the elimination diet on growth and nutrient intake in children with food protein induced gastrointestinal allergies. Clin Transl Allergy. 2016 Jul 14;6:25. doi: 10.1186/s13601-016-0115-x. eCollection 2016. PMID 27418957
- [Background] Mailhot G, Perrone V, Alos N, Dubois J, Delvin E, Paradis L, Des Roches A. Cow's Milk Allergy and Bone Mineral Density in Prepubertal Children. Pediatrics. 2016 May;137(5):e20151742. doi: 10.1542/peds.2015-1742. PMID 27244780
- [Background] Robbins KA, Wood RA, Keet CA. Milk allergy is associated with decreased growth in US children. J Allergy Clin Immunol. 2014 Dec;134(6):1466-1468.e6. doi: 10.1016/j.jaci.2014.08.037. Epub 2014 Oct 11. No abstract available. PMID 25312758
- [Background] Kim J, Kwon J, Noh G, Lee SS. The effects of elimination diet on nutritional status in subjects with atopic dermatitis. Nutr Res Pract. 2013 Dec;7(6):488-94. doi: 10.4162/nrp.2013.7.6.488. Epub 2013 Nov 29. PMID 24353835